CLINICAL TRIAL: NCT01438047
Title: OFDI in Dermatology
Brief Title: Optical Frequency Domain Imaging (OFDI) in Dermatology
Status: Withdrawn | Type: Observational
Why Stopped: The study was closed due to a shift in research priorities and a lack of resources available for the project.
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Benjamin Vakoc, Assistant Professor, Massachusetts General Hospital
Other Study IDs: 2010p001607
Record Dates: First submitted 2011-09-19; First posted 2011-09-21 (Estimated); Last update posted 2014-04-04 (Estimated); Status verified 2014-04

CONDITIONS: Port Wine Stain
Keywords: Port Wine Stain
MeSH Terms: conditions — Port-Wine Stain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a pilot exploratory study. The goal of this study is to evaluate a new imaging tool, optical frequency domain imaging (OFDI), to reveal the microvascular morphology of capillary malformations.

DETAILED DESCRIPTION:
The subject population will be composed of 8 subjects meeting the inclusion and exclusion criteria. Up to 8 subjects may be enrolled for the study after obtaining written, informed consent prior to participation in the study. Recruitment will be performed by direct advertisement to subjects inside and outside Brigham and Women's Hospital (BWH), including the BWH dermatology clinic. The study patients will be managed using standard of care in practice at the BWH dermatology clinic. The study will be conducted at Brigham and Women's Hospital Dermatology Clinic where the pulsed dye laser is housed.

Patients referred to the BWH dermatology clinic will be eligible for recruitment. The study nurse/staff involved in patient enrollment will be familiar with the care of this type of patients. The medical history of these patients will be examined to determine if the study eligibility requirements are met. If the patient is selected as a potential subject, a letter will be sent about 7 days prior to their scheduled exam to ask if they would care to participate. This time frame should allow time for the patient to consider study participation.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects: Fitzpatrick skin type I-VI, of either gender
2. Subjects must be between 18 and 80 years of age.
3. Subjects must have a not previously treated port wine stain of at least 1 cm2 on either a) trunk and extremities or b) face and neck.
4. Subjects are scheduled for PLD treatment of the port wine stain
5. Subjects must be willing and able to comply with all follow-up requirements.

Exclusion Criteria:

1. Subjects must not have active localized or systemic infections
2. Subjects must not be on aspirin.
3. Subjects must not be currently taking Accutane or be off Accutane for less than 6 months prior to initiation of the study.
4. Subjects must not be participating in potentially confounding research; e.g. a clinical study of any other unapproved investigational drug or device.
5. Subjects must not be pregnant or planning to become pregnant over the course of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing pulsed-dye laser for the treatment of capillary malformations at Brigham and Women's Hospital will be eligible for recruitment in this study.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-09; Primary Completion 2012-09 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
OFDI in Dermatology - Change from baseline in vascular density | 4 weeks
  There will be four times the patient is imaged using OFDI. Imaging is done to measure the vascular density within the specified area that is imaged. The first time imaging takes place is immediately prior to PDL treatment. The second in immediately following the treatment. The third and fourth imagings will be taken approximately four weeks after the initial visit. At this second visit the patient will have their second and final PDL treatment. An image will be take prior and following the PDL treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin J Vakoc, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- BWH, Boston, Massachusetts, United States